CLINICAL TRIAL: NCT06499558
Title: Suleyman Demirel University
Brief Title: Teaching Family Planning Skills With Standardized Patients"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, İlknur Atasever, Assistant Professor, Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: u3mjm2ey
Record Dates: First submitted 2024-05-23; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Educational Problems
Keywords: education; family planning; standard patient

STUDY DESIGN:
Intervention Model Description: In the study, participants are divided into two groups: the laboratory training group (the group receiving standard training) and the group receiving standard patient training.
Masking Description: In the study, participants are divided into two groups: the laboratory training group (the group receiving standard training) and the group receiving standard patient training. For this reason, blinding was not possible among the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Classical Training (Other): In the professional skills laboratory, students in the control group will practice family planning education skills
  Interventions: Other: Classical Training
- Standard Patient Interviews (Other): Students in the standard patient education group will receive standard patient education including a family planning counseling scenario.
  Interventions: Other: Standard Patient Interviews

INTERVENTIONS:
Other: Classical Training — Students in the education group will practice family planning education skills in the professional skills laboratory.
  Arms: Classical Training
Other: Standard Patient Interviews — Students in the standardized patient education group will receive training involving a family planning counseling scenario with standardized patients.
  Arms: Standard Patient Interviews

SUMMARY:
The research is planned to be carried out in the Simulated Patient Laboratory of Süleyman Demirel University Faculty of Medicine. The population of the research will consist of students taking the Hem 327 Women's Health and Diseases Nursing course in the fall semester of the 2023-2024 academic year (N: 179). Students receive training in small groups of 30-40 people in the professional skills laboratory. It is planned to study with a total of 80 students, 40 in the intervention group and 40 in the control group. Students will be assigned to intervention and control groups by lottery. The entire intervention and control group will receive theoretical training on "Family Planning", which is included in the 327 Women's Health and Diseases Nursing course. The course, conducted by the research faculty member using lecture, question-answer and discussion methods, will last three hours. Students participating in the study during the week of the theoretical course will be asked to fill out the Introductory Characteristics Form and the Family Planning Counseling Information Form.

DETAILED DESCRIPTION:
The main purpose of nursing education is; To train healthcare professionals who can combine theoretical knowledge with practice, and who have acquired critical thinking and effective problem-solving skills. Clinical practice is one of the most important elements of nursing teaching. It is thought that simulation training will be effective in preparing students for clinical practice and will increase their self-confidence in clinical practice by improving their clinical decision-making and application skills. Therefore, whether knowledge and skill gains can be transferred to nursing practice is an important area of interest in simulation research. The research is planned to be carried out in the Simulated Patient Laboratory of Süleyman Demirel University Faculty of Medicine. The population of the research will consist of students taking the Hem 327 Women's Health and Diseases Nursing course in the fall semester of the 2023-2024 academic year (N: 179). Students receive training in small groups of 30-40 people in the professional skills laboratory. It is planned to study with a total of 80 students, 40 in the intervention group and 40 in the control group. Students will be assigned to intervention and control groups by lottery. The entire intervention and control group will receive theoretical training on "Family Planning", which is included in the 327 Women's Health and Diseases Nursing course. The course, conducted by the research faculty member using lecture, question-answer and discussion methods, will last three hours. Students participating in the study during the week of the theoretical course will be asked to fill out the Introductory Characteristics Form and the Family Planning Counseling Information Form. In the same week, students in the control group will practice family planning education skills in the vocational skills laboratory. At the end of the application, students will fill out the Effective Communication Skills Evaluation Form and the Family Planning Education Skills Evaluation Form. Students in the intervention group are; They will participate in standard patient education that includes a family planning counseling scenario. Students will be given preliminary information before encountering a standard patient. During standard patient preparations; standard patients will be informed about the scenarios. Standard clothes and additional materials that patients will use while performing the scenario will be provided. Care will be taken to ensure that individuals serving as standard patients have previously taken part in other studies as standard patients. Then, the student will be brought together with the standard patient in the standard patient room of the clinical simulation training laboratory and a video recording will be taken at this time. The standard patient will behave in accordance with the patient role in the scenario given to him by the researcher. The application recording will be monitored by the researcher and the observer in the observation room in the standard patient room, and the Effective Communication Skills Evaluation Form and Family Planning Education Skill Evaluation Form will be filled in to evaluate the skill levels of the students. Then, a debriefing session will be held in the debriefing room, in line with the debriefing questions. Meanwhile, students will be given feedback on their deficiencies and performance in the application. Students' satisfaction and self-confidence towards this education will be evaluated with the Student Satisfaction and Self-Confidence Scale in Learning. The evaluation of the data will be done on a computer using the SPSS (Statistical Package For Social Sciences) 21.0 package program. In the analysis of data, percentage distributions, mean, standard deviation, chi-square test, and t-test in dependent groups will be used. Research findings will be evaluated at a 95% confidence interval and a significance level of p<0.05. In order to conduct the research, ethics committee approval was obtained from the Süleyman Demirel University Ethics Committee Presidency and legal permission was obtained from the Dean's Office of Süleyman Demirel University Faculty of Medicine, where the research will be conducted.

ELIGIBILITY:
Inclusion Criteria:

- To be a third-year nursing student at the Faculty of Health Sciences

• To consent to participate in the research.

Exclusion Criteria:

* Not completing any stage of the study
* Requesting to withdraw from the study
* Having previously taken the Obstetrics and Gynecology Nursing course

Ages: 21 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2024-05-31 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
Standard patient practice has an impact on students' satisfaction level. | through study completion, an average of 6 month
  Student Satisfaction and Confidence Scale in Learning

SECONDARY OUTCOMES:
The effect of standardized patient practice on students' self-confidence has been investigated | through study completion, an average of 6 month
  Family Planning Counseling Information Form, Effective Communication Form,Family Planning Education Skills Assessment Form

CONTACTS AND LOCATIONS:
Overall Officials: Ilknur Atasever, Assist. Prof., Principal Investigator — Suleyman Demirel University; Ilknur Atasever, Assist. Prof.., Principal Investigator — Suleyman Demirel University
Locations (1):
- Suleyman Demirel University Health Sciences Faculty Nursing Department, Isparta, Çünür, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Our plan aims to ensure transparent sharing of research results and accessibility to the scientific community. Individual participant data will be safeguarded in accordance with privacy standards.